CLINICAL TRIAL: NCT03330496
Title: Using Machine-learning Algorithms to Assess Acute Pain in Nonverbal Infants
Brief Title: Assessment of Pain in Newborns and Older Infants (Infant Pain Assessment Study =
Acronym: iPAS)
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Autonomous Healthcare, Inc. (Industry)
Responsible Party: Principal Investigator, Kanwaljeet Anand, Professor of Pediatrics, Anesthesiology, Perioperative & Pain Medicine, Stanford University
Other Study IDs: IRB-39076
Record Dates: First submitted 2017-10-24; First posted 2017-11-06 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Pain, Acute
Keywords: infant-newborn; infant-premature; pain; acute pain
MeSH Terms: conditions — Acute Pain; Premature Birth; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Preterm infants: preterm neonates (34-37 weeks gestational age, n=15)
  Interventions: Other: Pain Measurement
- Term infants: term newborns (37-42 weeks gestation, n=15)
  Interventions: Other: Pain Measurement
- Small infants: 1-3 month-old infants (n=15)
  Interventions: Other: Pain Measurement
- Older infants: 3-6 month-old infants (n=15)
  Interventions: Other: Pain Measurement

INTERVENTIONS:
Other: Pain Measurement — Measurement of infant responses (behavioral and physiological) during a painful procedure.

SUMMARY:
Pain assessments in non-verbal, critically ill infants represent an important clinical challenge. Older children or adults can easily express their pain, but infants lack that capability. They frequently experience repetitive acute pain during routine ICU care, but their analgesic management flounders on the horns of a dilemma: (a) failure to treat infant pain leads to immediate clinical instability and potentially long-term physical, behavioral, and cognitive sequelae, vs. (b) strong analgesics may increase risks for medical complications and/or impaired brain growth. Bedside nurses currently assess pain using pain scores, before taking action to ameliorate pain. Pain scores increase nursing workload and provide subjective assessments, rather than objective data for evaluating infant pain. Consequently, infants exposed to skin-breaking procedures, surgery, or other painful conditions often receive variable and inconsistent pain management in the ICU. The investigators aim to develop a multimodal pain assessment system, using sensor fusion and novel machine learning algorithms to provide an objective measure of pain that is context-dependent and rater-independent. This will enhance the quality of pain management in ICUs and allow continuous pain monitoring in real-time.

ELIGIBILITY:
Inclusion Criteria:

* 1. All infants less than 6 months of corrected chronological age. 2. Infants admitted to the participating ICUs at LPCH (NICU, PICU, CVICU). 3. Require an acute painful procedure for routine clinical care.

Exclusion Criteria:

1. Newborns with birth trauma, intrapartum asphyxia (5-minute Apgar Score <4 or cord pH < 7.01), fetal growth restriction (birth weight < 5th percentile for gestation), congenital anomalies or metabolic disorders, or any kind of brain injury.
2. Newborns born to mothers with a history of heavy smoking or drug abuse (alcohol, cocaine, ketamine, heroin/other opiates) or psychiatric drugs used during this pregnancy.
3. Newborns and infants requiring positive pressure ventilation using a face mask (BiPAP) or endotracheal tube (conventional or high-frequency ventilators).
4. Newborns and infants receiving continuous infusions of opioid drugs (morphine, fentanyl, others) and nerve blocks or neuraxial analgesia affecting the site of the invasive procedure during the 24 hours prior to study entry. (Note: Infants receiving intermittent opioids or non-opioid analgesics (acetaminophen, ibuprofen, ketorolac, others) WILL NOT be excluded).
5. Newborns and infants with facial anomalies, injuries or other pathologies affecting the facial area.

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We will collect data from 30 study subjects in each of the following age groups:
  * Preterm infants (34-37 weeks, postnatal age 3-30 days)
  * Term newborns (37-42 weeks gestation, less than 1 month of age)
  * Infants from 1-3 months age, and
  * Older infants from 3-6 months age. A total of 120 subjects will be recruited before study closure.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Pain Measurement (all infants) | 10 minutes
  Visual Analogue Scale (VAS) measures pain intensity based on observer assessment on a scale from 1 to 10, where higher values indicate more intense pain.

SECONDARY OUTCOMES:
Pain Measurement | 30 minutes
  Facial Expressions specific for infant pain will be assessed, including nasolabial furrow and brow bulge. Presence or absence as well as the duration for each facial expression will be recorded during the painful procedure. These facial expressions were chosen from the Neonatal Facial Coding Scale (NFCS) and the Premature Infant Pain Profile (PIPP).
Pain Measurement (newborns 0-30 days) | 5 minutes
  Neonatal Pain, Agitation and Sedation Scale (N-PASS) measures level of sedation versus increasing pain or agitation in newborns. Scores range from -10 to +10, where negative scores denote increasing levels of sedation, zero indicates a neutral condition, and positive scores indicate increasing pain intensity and/or agitation.
Pain Measurement (newborns 0-30 days) | 8 minutes
  Premature Infant Pain Profile - Revised (PIPP-R) measures pain intensity in newborns, with scores ranging from 0 to 21, higher scores indicating greater pain (adjusted for prematurity and behavioral state).
Pain Measurement (infants 1-6 months) | 3 minutes
  Face, Legs, Activity, Cry, Consolability scale (FLACC scale) measures pain in children between the ages of 2 months and 7 years. The scale is scored in a range of 0-10 with 0 representing no pain and 10 indicating severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Kanwaljeet S Anand, MBBS, D.Phil., Principal Investigator — Prof.
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared

REFERENCES:
- [Derived] Roue JM, Avnit A, Gholami B, Haddad WM, Anand KJS. Objective Detection of Newborn Infant Acute Procedural Pain Using EEG and Machine Learning Algorithms. Paediatr Neonatal Pain. 2025 Mar 10;7(1):e70001. doi: 10.1002/pne2.70001. eCollection 2025 Mar. PMID 40066435
- [Derived] Roue JM, Morag I, Haddad WM, Gholami B, Anand KJS. Using sensor-fusion and machine-learning algorithms to assess acute pain in non-verbal infants: a study protocol. BMJ Open. 2021 Jan 6;11(1):e039292. doi: 10.1136/bmjopen-2020-039292. PMID 33408199